CLINICAL TRIAL: NCT01378819
Title: Three Ports Placed in the Line Alba of the Abdomen (3-midline-ports Technique): an Alternative Approach for Laparoscopic Cholecystectomy
Brief Title: 3-midline-ports Cholecystectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Jaime Ruiz-Tovar, Hospital General de Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMH
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2010-02

CONDITIONS: Postoperative Pain
Keywords: laparoscopic cholecystectomy; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: 3-midline-ports laparoscopic cholecystectomy — The laparoscopic cholecystectomy will be performed through 3 ports placed in the line alba.
Procedure: 3-midline-ports laparoscopic cholecystectomy — Laparoscopic cholecystectomy will be performed through 3 ports placed in the line alba.

SUMMARY:
The 3-midline-ports technique is a safety approach and associates lower postoperative pain, when compared with the standard "French" technique.

DETAILED DESCRIPTION:
The patients will be randomized into 2 groups: those patients undergoing laparoscopic cholecystectomy following the "French" technique (Group 1) and those ones undergoing the 3-midline-ports approach (Group 2).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cholecystectomy for symptomatic gallstones.

Exclusion Criteria:

* Diagnosis of acute cholecystitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours
  The postoperative pain will be investigated 24 hours after surgery